CLINICAL TRIAL: NCT02807233
Title: Observational, Multicenter, Cross-sectional, Observational Study to Evaluate the Effectiveness in Routine Clinical Practice of Lanreotide Autogel 120 mg at Extended Dosing Intervals (>4 Weeks) for the Treatment of Acromegaly: SOMACROL Study.
Brief Title: Lanreotide Autogel 120 mg at Extended Dosing Intervals (>4 Weeks) in Acromegalic Subjects
Acronym: SOMACROL
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-ES-52030-352; IPS-SOM-2015-01 (Other: Spanish Drug Agency AEMPS)
Record Dates: First submitted 2016-05-27; First posted 2016-06-21 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the effectiveness in IGF-1 control of lanreotide Autogel (ATG) 120 mg at extended dosing intervals (EDIs) (>4 weeks) in subjects with acromegaly in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥ 18 years
* Diagnosed with acromegaly
* Receiving treatment with ATG 120 mg at extended dosing intervals (> 4 weeks) for at least six months before the study visit.
* Assay data (blood GH and IGF-1 levels) from immediately before the study visit (performed at least six months after starting the treatment) is available.
* Able to sign the informed consent form for study participation.

Exclusion Criteria:

* Received radiation therapy treatment in the last six months.
* Active participation in another clinical study.
* Physical or mental disorders that, in the investigator's opinion, could affect their ability to sign the informed consent form.
* Pregnancy or breastfeeding for female patients.
* No data in their medical records on the treatment start date for ATG 120 mg at extended dosing intervals or on changes to the schedule of administration over the last six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with a normal Insulin-like Growth Factor 1 (IGF-1) level in the assay before the study visit. | Day 1

SECONDARY OUTCOMES:
Percentage of subjects with Growth hormone (GH) levels ≤ 2.5 ng/mL or ≤ 1 ng/mL in the assay before the study visit. | Day 1
Percentage of subjects treated with lanreotide autogel (ATG) 120 mg for ≥ 6 months with dosing intervals of five, six, seven or eight weeks. | Day 1
Percentage of subjects whose dosing regimen has been changed in the six months before the study. | Day 1
Preference for self-administered injections or administration in an outpatient clinic by a medical professional. | Day 1
Acromegaly Quality of Life Questionnaire (AcroQoL) in subjects after ≥ 5 months of treatment with ATG 120 mg at extended dosing intervals. | Day 1
  Total score and score per domain
EuroQol-5D (EQ-5D) questionnaire in subjects after ≥ 5 months of treatment with ATG 120 mg at extended dosing intervals. | Day 1
  Total score and score per domain
Treatment Satisfaction Questionnaire for Medication-9 (TSMQ-9) in subjects treated with ATG 120 mg at extended dosing intervals after ≥ 5 months. | Day 1
  Total score and score per domain
Variations between theoretical and real treatment compliance for non-medical reasons. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (39):
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Sao Jöao, Porto
- Spain (37):
  - Hospital Univ. Nuestra Sra. Candelaria, Santa Cruz, Tenerife
  - Complejo Hospitalario Univ. A Coruña, A Coruña
  - Hospital Univ. Príncipe de Asturias, Alcalá de Henares
  - Hospital General Univ. de Alicante, Alicante
  - Hospital Univ. La Ribera, Alzira
  - Hospital Infanta Cristina, Badajoz
  - Hospital Cruces, Barakaldo
  - Hospital Puerta del Mar, Cadiz
  - Hospital Ciudad Real, Ciudad Real
  - Hospital Reina Sofía, Córdoba
  - Hospital de Getafe, Getafe
  - Hospital Univ. Girona Dr. Josep Trueta, Girona
  - Hospital de Jaén, Jaén
  - Hospital Bellvitge, L'Hospitalet de Llobregat
  - Hospital Univ. León, León
  - Hospital Arnau de Vilanova, Lleida
  - Hospital La Princesa, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital La Paz, Madrid
  - Hospital Univv. La Paz, Madrid
  - Hospital Puerta del Hierro, Madrid
  - Hospital Civil de Málaga, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Univ. Central de Asturias, Oviedo
  - Hospital Univ. Son Espases, Palma
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Infanta Sofía, San Sebastián de los Reyes
  - Hospital Clínico Univ. Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital Univ. Alava, Terrassa
  - Hospital Univ. Mutua de Terrassa, Terrassa
  - Hospital Obispo Polanco, Teruel
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico de Valencia, Valencia
  - Hospital Univ. La Fe, Valencia
  - Hospital Clínico Univ. Valladolid, Valladolid
  - Hospital Miguel Servet, Zaragoza